CLINICAL TRIAL: NCT05250609
Title: Clinical and Radiographic Evaluation of Resin Endocrown as Long Term Interim Restoration Versus Stainless Steel Crown for Endodontically Treated First Permanent Molar in Children: Randomized Controlled Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basheer Ali Mabkhot, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422021510951
Record Dates: First submitted 2022-02-05; First posted 2022-02-22 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The statistician will be blinded throughout the whole procedures (double blind). Principle investigator will be responsible for all clinical procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Endocrown "composite". (Experimental): Composite Endocrown will be used as an extra-coronal restoration in endodontically treated mutilated first permanent molar
  Interventions: Other: Endocrown "composite".
- Comparator / Control: Stainless steel crown. (No Intervention): Stainless steel crown will be used as an extra-coronal restoration in endodontically treated mutilated first permanent molar

INTERVENTIONS:
Other: Endocrown "composite". — It is a type of restoration has been shown a great success in adult and recently has been suggested for children
  Arms: Intervention: Endocrown "composite".

SUMMARY:
management of endodontically treated first permanent molar with deep dental caries is one of the challenging procedure that the operator face. Using resin endocrown or stainless steel crown restoration to make comparison which one is more successful in children.

DETAILED DESCRIPTION:
Diagnostic procedure:

Diagnosis of the cases will be performed according to guidelines of AAPD 2017 for treatment of irreversible pulpitis and necrotic pulp therapy in mandibular first permanent molar . Preoperative periapical radiograph will be taken

Intra operative procedure:

Local anaesthesia administration using articaine 4% with epinephrine 1:100000. Rubber dam application and access cavity preparation will be established using a sterile bur. Root Canal Treatment will be done and then the dental orifices of the pulp chamber will be sealed using a flowable composite.

The immediate postoperative radiograph will be done to reveal optimal root canal treatment.

In the intervention group:

The preparation of cavity design will be as following:

Preparation of occlusal surface will be done with wheel stone to create 2 mm occlusal clearance; the occlusal surface will be prepared flat to create a butt-joint. The junction between the occlusal and mesial cavity will be rounded to produce cervical side walk. • Divergence of the inner cavity walls will be obtained using a tapered stone with a rounded end (TR- Dia Bur Mani).

Impression will be taken for the prepared tooth structure using addition silicone material (Elite HD Zermach, Italy), stone model will be poured for fabrication of endocrown to allow for blockage of any undercuts in the pulp chamber cavity. Finished final endocrown restoration will be cemented in place using self-adhesive universal dual cured resin cement (rely X Unicem, 3M, USA).

In the control group tooth preparation will be made as follow:

By reducing mesial, distal and occlusal surface. The crown margin will be placed just apically to the gingival margin and carefully adjusted to give an accurate fit in this region. The crown will be cemented with glass ionomer cement.

Follow up:

Clinical and evaluation will be performed at 1 st week, 3, 6, 9 and 12 months. Radiograph evaluation will be performed at, 1 st week, 6 and 12 months

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children in age range from 10 to 13 years

  * Mandibular first permanent molar indicated for root canal treatment with closed apex.
  * Presence of at least two to three sound walls of tooth.
  * Absence of internal or external pathologic root resorption.
  * Normal occlusion without any para-functional habits.
  * Parent or guardian agree for participant in the study

Exclusion Criteria:

* Excessive mobility.
* Children with underlying systemic disease.
* Children with special health care needs.
* Poor oral hygiene.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | one year
  Will be recorded by using modified wong-baker pain scale (0 -3). Zero= no pain, 1= slight pain, 2=moderate pain, 3= severe pain. Principle investigator will ask the patient about the pain.
Gingival bleeding | one year
  Gingival Index(GI)Scale (0-3): score 0: normal gingiva, score1: mild inflammation, slight change in colour, slight oedema, no bleeding on probing, score2: moderate inflammation, redness, oedema, and glazing, bleeding on probing, score3: severe inflammation, marked redness and oedema, ulceration tendency to spontaneous bleeding.
Retention | one year
  Clinical evaluation by Principle investigator. Binary (Yes/No)
Patient satisfaction | one year
  Patient and guardian satisfaction with restorative treatment was classified as (score from 1-4) 1= very dissatisfied, 2= dissatisfied, 3= satisfied and 4= very satisfied
Probing pocket depth (PPD) | one year
  Periodontal probe. (1-5 mm):It will be measured in mesiobuccal, distobuccal, mesiolingual, and distolingual areas. The periodontal probe will be inserted into the gingival sulcus parallel to the longitudinal axis of the tooth and will be moved in a walking fashion.

SECONDARY OUTCOMES:
Radiograph in Terms of root fracture | one year
  Digital radiographic Evaluation. Binary(Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Basheer MAbkhot, Cairo, Jiza, Egypt

REFERENCES:
- [Derived] Mabkhot BA, Taha SEE, Sabry SM. Clinical and radiographic assessment of composite CAD/CAM endocrowns and stainless steel crowns for endodontically treated first permanent molars in Egyptian children: randomized controlled pilot study. BMC Oral Health. 2025 May 31;25(1):864. doi: 10.1186/s12903-025-06192-y. PMID 40450229